CLINICAL TRIAL: NCT06253728
Title: Comprehensive Study of Biochemical Response to Alternative Protein Sources in Different Food Matrices
Brief Title: A Study of Biochemical Response to Alternative Proteins
Acronym: COBRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: A80406
Record Dates: First submitted 2024-01-30; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Postprandial Hyperglycemia; Overweight and Obesity; Type2diabetes
MeSH Terms: conditions — Hyperglycemia; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Meal 1 (Experimental): Meal with plant protein and fiber in an intact structure
  Interventions: Dietary Supplement: High fiber and protein meal
- Meal 2 (Experimental): Meal with plant protein and fiber, where the cell structure is broken
  Interventions: Dietary Supplement: High fiber and protein meal
- Meal 3 (Placebo Comparator): Low protein and low fiber cereal
  Interventions: Dietary Supplement: Control
- Meal 4 (Experimental): High protein and low carbohydrate bread with animal proteins
  Interventions: Dietary Supplement: High fiber and protein meal
- Meal 5 (Experimental): High protein and low carbohydrate bread with plant protein
  Interventions: Dietary Supplement: High fiber and protein meal

INTERVENTIONS:
Dietary Supplement: High fiber and protein meal — In the intervention participants are assigned to eat high protein and fiber meal that differ in protein source or structure.
  Arms: Meal 1; Meal 2; Meal 4; Meal 5
Dietary Supplement: Control — The control meal is low fiber and low protein meal.
  Arms: Meal 3

SUMMARY:
The overall objective of this research is to determine the digestive faith and health impact of protein and fiber rich foods in different food matrices in type 2 diabetes risk population. This is achieved by controlled postprandial intervention where plasma amino acids, lipids, glucose metabolism, bile acids and microbial metabolites are evaluated as well as fecal microbiota and metabolites.

DETAILED DESCRIPTION:
Detailed research aim of this controlled, randomized crossover postprandial clinical study are:

1. To study the impact of complex plant- and animal-based foods on glucose metabolism, acute inflammation, and markers of microbial fermentation of fiber and proteins.
2. To investigate the difference in the gut mediated metabolism induced by naturally occurring fiber fraction bound plant protein or by plant protein with added fiber when compared to animal protein.
3. To conduct in vitro experiments using fecal samples from participants in the meal study to investigate the distinctions between different animal and plant proteins on both host and microbial metabolites, as well as the function of the gut barrier.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years of age
* BMI >25 kg/m2 and <35 kg/m2
* Waist circumference with females >85 cm and with males >100 cm

Exclusion Criteria:

* Certain chronic diseases requiring regular medication (e.g., type 2 diabetes, chronic liver, kidney, thyroid, or gastrointestinal diseases)
* Pregnancy or breastfeeding
* Gluten-free or vegan diet
* Use of antibiotics within the last 12 months
* Gastrointestinal surgery within the last two years
* High alcohol consumption

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-06-03 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma amino acids | 0-4 hours
  Plasma free amino acids were measured at 0, 30, 60, 90, 180, and 240 minutes after consuming the study meal.
Gut derived metabolites | 0-24 hours
  Gut derived metabolites are measured with untargeted metabolomics from plasma at 12 hours after consuming the study meal. From fecal sample, the metabolomics are measured at 24 hours after consuming the study meal. Plasma short chain fatty acids are quantified at 12 hours after consuming the study meal.

SECONDARY OUTCOMES:
Plasma glucose | 0-4 hours
  Plasma glucose is measured at 0, 30, 60, 90, 180, and 240 minutes after consuming the study meal.
Inflammation marker | 0-4 hours
  Plasma IL-22 is measured at 0, 60, 240 minutes after consuming the study meal.
Plasma triglycerides | 0-4 hours
  Plasma triglycerides are measured at 0, 30, 60, 90, 180, and 240 minutes after consuming the study meal.
Urine para-cresol | 24 hours
  The amount of para-cresol is measured from urine sample at 24 hours after consuming the study meal.
Plasma insulin | 0-4 hours
  Plasma insulin is measured at 0, 30, 60, 90, 180, and 240 minutes after consuming the study meal.
Plasma free fatty acids | 0-4 hours
  Plasma free fatty acids are measured at 0, 30, 60, 90, 180, and 240 minutes after consuming the study meal.

CONTACTS AND LOCATIONS:
Overall Officials: Marjukka Kolehmainen, Professor, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No